CLINICAL TRIAL: NCT06570785
Title: Contralateral Limb Cannulation Using Intra-Operative Positioning SystemTechnology in Endovascular Aneurysm Repair
Brief Title: IOPS Technology During Cannnulation of Contralateral Limb in EVAR
Acronym: IOPS
Status: Not yet recruiting | Type: Observational
Sponsor: Clinical Centre of Serbia (Other)
Collaborators: Centerline Biomedical, Inc. (Industry)
Responsible Party: Principal Investigator, Petar Zlatanovic, Principal Investigator MD PhD FEBVS, Clinical Centre of Serbia
Other Study IDs: IOPS study
Record Dates: First submitted 2024-08-21; First posted 2024-08-26 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Abdominal Aortic Aneurysm; Abdominal Aortic Aneurysm Without Rupture; Radiation Exposure
Keywords: Abdominal Aortic Aneurysm; EndoVascular Aneurysm Repair; Radiation Protection
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- IOPS group: Patients with AAA undergoing standard EVAR according to the IFU using IOPS technology for visulisation of guidewires and catheter for the cannulation of contralateral limb.
  Interventions: Device: Intra-Operative Positioning System (IOPS)
- Conventional group: Patients with AAA undergoing standard EVAR according to the IFU using standardised approach and materials.
  Interventions: Device: Conventional group

INTERVENTIONS:
Device: Intra-Operative Positioning System (IOPS) — This medical device provides surgeons with 3D visualization for increased surgical precision while reducing the use of contrast dye and radiation exposure for patients and healthcare professionals alike. IOPS provides 3D electromagnetic navigation of interventional devices as an adjunct to fluoroscopy. During the intervention, the IOPS devices can be visualized with on-screen image guidance. The console is operated by a technician under a physician's instruction. The IOPS guidewires and catheters can be used together or combined with off-the-shelf 0.035-inch catheters and guidewires, as needed.
  Groups: IOPS group
Device: Conventional group — This group will be treated using standardised materials (wires, catheters) during EVAR.
  Groups: Conventional group

SUMMARY:
Short-term results are favorable for EndoVascular Aneurysm Repair (EVAR) compared to open surgery. One of the major drawbacks to this shift is the need for fluoroscopy and contrast dyes to visualise endovascular devices. The use of fluoroscopy exposes both patients and caregivers to harmful ionizing radiation. Because of the harmful effects of radiation, recent radiation protection guidelines strongly recommend as low as reasonably achievable (ALARA) principle. The need for additional radiation-reducing navigation techniques is high, with the ultimate goal of performing endovascular procedures without radiation at all.

In response to these challenges, Centerline Biomedical (Cleveland, Ohio, USA) has developed a proprietary electromagnetic tracking and positioning system called the Intra-Operative Positioning System (IOPS). This medical device provides surgeons with 3D visualization for increased surgical precision while reducing the radiation exposure for patients and healthcare professionals. IOPS provides 3D electromagnetic navigation of interventional devices as an adjunct to fluoroscopy. During the intervention, the IOPS devices can be visualized with on-screen image guidance. The IOPS guidewires and catheters can be used together or combined with off-the-shelf 0.035-inch catheters and guidewires, as needed.

This study aims to describe the influence of IOPS technology on radiation exposure during cannulation of the contralateral limb (CL) during standard EVAR.

DETAILED DESCRIPTION:
Background:

The current standard of care for abdominal aortic aneurysm (AAA) is endovascular aneurysm repair (EVAR) which has been suggested as the treatment of choice by both European and American guidelines . Although short-term results are favorable for EVAR compared to open surgery, one of the major drawbacks to this shift is the need for fluoroscopy and contrast dyes to visualise endovascular devices. The contrast dyes used during these procedures can induce renal failure in patients with preexisting renal dysfunction. Meanwhile, the use of fluoroscopy exposes both patients and caregivers to harmful ionizing radiation. Because of the harmful effects of radiation, recent radiation protection guidelines strongly recommend as low as reasonably achievable (ALARA) principle.

In response to these challenges, Centerline Biomedical (Cleveland, Ohio, USA) has developed a proprietary electromagnetic tracking and positioning system called the Intra-Operative Positioning System (IOPS). This medical device provides surgeons with 3D visualization for increased surgical precision while reducing the use of contrast dye and radiation exposure for patients and healthcare professionals alike. IOPS provides 3D electromagnetic navigation of interventional devices as an adjunct to fluoroscopy. Image guidance is provided using 3D maps of the vasculature, generated from thin-slice contrast-enhanced preoperative computerised tomography angiography (CTA). At the start of the procedure, a self-adhesive sterile fiducial tracking pad is attached to the patient's lumbar region, and the angiography system is used to perform a non-contrast-enhanced cone-beam CT scan. The cone beam CT volume is then loaded onto the IOPS cart and manually aligned with the preoperative CT volume. This work can be performed in parallel with achieving vascular access, with minimal effects on the procedure time. During the intervention, the IOPS devices can be visualized with on-screen image guidance. The console is operated by a technician under a physician's instruction. The IOPS guidewires and catheters can be used together or combined with off-the-shelf 0.035-inch catheters and guidewires, as needed. This technology has been used by other centres for visceral and renal cannulation during complex aortic aneurysm procedures.

Previously there have been publications on the use of Fiber Optic Real Shape (FORS) Technology with both complex and standard endovascular aneurysm repair (EVAR) showing the potential benefit of this technology in procedural time and radiation reduction. However, the need for additional radiation-reducing navigation techniques is high, with the ultimate goal of performing endovascular procedures without radiation at all.

This study aims to describe the influence of IOPS technology on radiation exposure during cannulation of the contralateral limb (CL) during standard EVAR.

Study outcome and sample size:

Technical success of using IOPS technology during cannulation of CL Navigation time expressed through total procedural time, CL cannulation time, fluoroscopy time (overall and during CL cannulation) Radiation exposure parameters that were described in the latest European Society for Vascular Surgery (ESVS) radiation guidelines: cumulative air kerma (CAK), kerma area product (KAP), fluoroscopy time (FT) (4) To ensure sufficient statistical power to answer hypothetical questions, 80 subjects will be entered into the database. Navigation time and radiation exposure parameters are used to calculate the sample size. Assuming the difference in terms of both parameters, 30 patients are required in each arm to achieve a statistical power of 85% at p=0.05. With two arms (conventional and IOPS group), assuming a 20% rate of missing data, a total N of 80 patients is required.

Research Design:

This prospective study includes patients with standard AAA undergoing EVAR within instructions for use (IFU) treated from September 1st, 2024 until May 1st, 2025 at the Clinic for Vascular and Endovascular Surgery, University Clinical Centre of Serbia.

Procedures Involved:

This study will not impact the care that patients receive. Patient data will be compiled and analyzed to accomplish the proposed study objectives. Data collection will include demographic information, patient-related factors, comorbidities, diagnostic imaging information (describing the morphology of the aortoiliac segment), and periprocedural information related to the timing and radiation.

Data management:

After the data has been collected at a participating institution, the data will be transmitted to an online database which will be available only to a central analytic center located at the Clinic for Vascular and Endovascular Surgery/University Clinical Center of Serbia/Medical Faculty, University of Belgrade.

Risks to Subjects:

As this is a prospective observational study performing EVAR in standard AAA using new radiation protection technology for visualisation of wires and catheters in a newly equipped angio suite, there are minimal potential physical risks to subjects. There is also a minimal risk of breach of confidentiality that could occur when patient information is collected and analyzed for the proposed study. However, appropriate measures will be taken to minimize the risk as much as possible. All information recorded will be de-identified. This study will abide by all regulations related to protecting human subjects and protected health information.

Potential Benefits to Subjects:

There is a potential benefit to the subjects involved in the IOPS group. Hypothetically they will have lower procedural times and lower radiation doses during CL cannulation. Future patients treated with this technology might have reduced radiation and cannulation times. This will make it possible to perform more and more procedures with a minimal amount of radiation, or even without radiation at all.

Statistics and Data Analysis:

Continuous variables will be described using the median and interquartile range or mean and standard deviation. Categorical variables will be described using frequencies and percentages. Group comparisons will be performed by using the Student t-test or Mann-Whitney U test, as appropriate. Categorical data will be expressed as percentages and will be compared using the chi-square test or Fisher exact test. Differences will be considered statistically significant at p < 0.05. Analyses will be performed using SPSS software, version 28.0 (SPSS, Chicago, ILLINOIS, USA).

Conflict of Interest:

Since this is a physician-initiated trial, the investigators have no conflict of interest to report.

Funding Source:

There are no plans to apply for additional grants or additional funding. No funding is required for the completion of this study.

Publication Plan:

All research personnel included in this project will be eligible for authorship in any resulting abstracts and publications following the qualifications outlined by the International Committee of Medical Journal Editors. The order of authors will be determined prior to manuscript development and depend on each individual's contribution to the study.

ELIGIBILITY:
Inclusion Criteria:

- All patients (over 18 years of age) with infrarenal AAA treated between 1st September 2024 and 1st May 2025 undergoing standard EVAR according to the IFU

Exclusion Criteria:

* Patients who are pregnant
* Patients who are under 40 years of age
* Patients who have symptomatic or ruptured AAA
* Patients with more advanced AAA: juxtarenal, pararenal, suprarenal, thoracic, thoracoabdominal AAA
* Non-atherosclerotic origin of disease: dissection, connective tissue disorders, mycotic AAA, posttraumatic AAA
* Patients who were treated in a conservative manner
* Patients undergoing open surgery
* Patients undergoing more advanced treatment options: fenestrated/branched EVAR, endostaplers, chimney EVAR, iliac branch devices, etc.

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with infrarenal AAA undergoing standard EVAR according to the IFUs of the manufacturer will be stratified into two groups:
  1. IOPS group (used during CL cannulation)
  2. Conventional group (as usual using a standardised approach for EVAR)
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-01-20 (Estimated); Primary Completion 2025-09-08 (Estimated); Study Completion 2025-11-03 (Estimated)

PRIMARY OUTCOMES:
Fluoroscopic time per participant required for cannulation | Cannulation of contralateral limb during the intervention
  Record cumulative fluoroscopy time reported by fluoroscopic system before and after cannulation of contralateral limb
Number of participants with technical success of gate catheterisation | Cannulation of contralateral limb during the intervention
  Definition of technical success with fluoroscopy: Cannulation completed retrograde; Definition of technical success with IOPS: Cannulation completed retrograde using IOPS catheter

SECONDARY OUTCOMES:
Clock time per participant required for cannulation | Cannulation of contralateral limb during the intervention
  Use stopwatch, or record clock time before and after cannulation of contralateral limb
Radiation dose per participant during cannulation | Record radiation reported by fluoro system before and after cannulation of contralateral limb during the intervention
  Cumulative air kerma [CAK], air kerma area product [KAP], excluding digital subtraction angiography time

CONTACTS AND LOCATIONS:
Overall Officials: Igor Koncar, MD PhD, Study Chair — University Clinical Centre of Serbia
Locations (1):
- Clinical Center of Serbia, Belgrade, Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: Undecided
This will be decided among the study group, once study has been completed.

REFERENCES:
- [Background] Wanhainen A, Van Herzeele I, Bastos Goncalves F, Bellmunt Montoya S, Berard X, Boyle JR, D'Oria M, Prendes CF, Karkos CD, Kazimierczak A, Koelemay MJW, Kolbel T, Mani K, Melissano G, Powell JT, Trimarchi S, Tsilimparis N; ESVS Guidelines Committee; Antoniou GA, Bjorck M, Coscas R, Dias NV, Kolh P, Lepidi S, Mees BME, Resch TA, Ricco JB, Tulamo R, Twine CP; Document Reviewers; Branzan D, Cheng SWK, Dalman RL, Dick F, Golledge J, Haulon S, van Herwaarden JA, Ilic NS, Jawien A, Mastracci TM, Oderich GS, Verzini F, Yeung KK. Editor's Choice -- European Society for Vascular Surgery (ESVS) 2024 Clinical Practice Guidelines on the Management of Abdominal Aorto-Iliac Artery Aneurysms. Eur J Vasc Endovasc Surg. 2024 Feb;67(2):192-331. doi: 10.1016/j.ejvs.2023.11.002. Epub 2024 Jan 23. PMID 38307694
- [Background] Chaikof EL, Dalman RL, Eskandari MK, Jackson BM, Lee WA, Mansour MA, Mastracci TM, Mell M, Murad MH, Nguyen LL, Oderich GS, Patel MS, Schermerhorn ML, Starnes BW. The Society for Vascular Surgery practice guidelines on the care of patients with an abdominal aortic aneurysm. J Vasc Surg. 2018 Jan;67(1):2-77.e2. doi: 10.1016/j.jvs.2017.10.044. PMID 29268916
- [Background] Antoniou GA, Antoniou SA, Torella F. Editor's Choice - Endovascular vs. Open Repair for Abdominal Aortic Aneurysm: Systematic Review and Meta-analysis of Updated Peri-operative and Long Term Data of Randomised Controlled Trials. Eur J Vasc Endovasc Surg. 2020 Mar;59(3):385-397. doi: 10.1016/j.ejvs.2019.11.030. Epub 2019 Dec 30. PMID 31899100
- [Background] Zlatanovic P, Davidovic L, Mascia D, Ancetti S, Yeung KK, Jongkind V, Viitala H, Venermo M, Wiersema A, Chiesa R, Gargiulo M. Acute kidney injury in patients undergoing endovascular or open repair of juxtarenal or pararenal aortic aneurysms. J Vasc Surg. 2024 Jun;79(6):1347-1359.e3. doi: 10.1016/j.jvs.2024.02.021. Epub 2024 Feb 22. PMID 38395093
- [Background] Modarai B, Haulon S, Ainsbury E, Bockler D, Vano-Carruana E, Dawson J, Farber M, Van Herzeele I, Hertault A, van Herwaarden J, Patel A, Wanhainen A, Weiss S, Esvs Guidelines Committee, Bastos Goncalves F, Bjorck M, Chakfe N, de Borst GJ, Coscas R, Dias NV, Dick F, Hinchliffe RJ, Kakkos SK, Koncar IB, Kolh P, Lindholt JS, Trimarchi S, Tulamo R, Twine CP, Vermassen F, Document Reviewers, Bacher K, Brountzos E, Fanelli F, Fidalgo Domingos LA, Gargiulo M, Mani K, Mastracci TM, Maurel B, Morgan RA, Schneider P. Editor's Choice - European Society for Vascular Surgery (ESVS) 2023 Clinical Practice Guidelines on Radiation Safety. Eur J Vasc Endovasc Surg. 2023 Feb;65(2):171-222. doi: 10.1016/j.ejvs.2022.09.005. Epub 2022 Sep 18. No abstract available. PMID 36130680
- [Background] Finnesgard EJ, Simons JP, Jones DW, Judelson DR, Aiello FA, Boitano LT, Sorensen CM, Nguyen TT, Schanzer A. Initial single-center experience using Fiber Optic RealShape guidance in complex endovascular aortic repair. J Vasc Surg. 2023 Apr;77(4):975-981. doi: 10.1016/j.jvs.2022.11.041. Epub 2022 Nov 13. PMID 36384183
- [Background] Klaassen J, Hazenberg CEVB, Bloemert-Tuin T, Wulms SCA, Teraa M, van Herwaarden JA. Editor's Choice - Radiation Dose Reduction During Contralateral Limb Cannulation Using Fiber Optic RealShape Technology in Endovascular Aneurysm Repair. Eur J Vasc Endovasc Surg. 2024 Apr;67(4):594-600. doi: 10.1016/j.ejvs.2023.10.041. Epub 2023 Nov 3. PMID 37925100
- [Background] Muluk SC, Elrakhawy M, Chess B, Rosales C, Goel V. Successful endovascular treatment of severe chronic mesenteric ischemia facilitated by intraoperative positioning system image guidance. J Vasc Surg Cases Innov Tech. 2021 Nov 22;8(1):60-65. doi: 10.1016/j.jvscit.2021.11.001. eCollection 2022 Mar. PMID 35118217
- See also: Link to the further description of IOPS technology — https://centerlinebiomedical.com/